CLINICAL TRIAL: NCT02658058
Title: A Randomized Controlled Trial of Pre-procedural Ultrasound Techniques Versus the Conventional Landmark Technique of Spinal Anesthesia in Elderly Patients
Brief Title: Pre-procedural Ultrasound Techniques Versus Conventional Landmark Technique of Spinal Anesthesia in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Sahar Sayyid, MD, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ANES.SS.13
Record Dates: First submitted 2015-11-11; First posted 2016-01-18 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Anesthesia
Keywords: Ultrasound; Spinal anesthesia; Elderly; Landmark

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Landmark technique (Active Comparator): As intervention, patients in this group are administered landmark guided midline spinal anesthesia.
  Interventions: Other: Landmark technique
- Ultrasound-guided paramedian technique (Experimental): As intervention, patients in this group are administered spinal anesthesia based on preprocedural ultrasound-guided paramedian technique using parasagittal oblique view
  Interventions: Other: Ultrasound-guided paramedian technique
- Ultrasound-guided midline technique (Experimental): As intervention, patients in this group are administered spinal anesthesia based on preprocedural ultrasound-guided midline technique using transverse median view
  Interventions: Other: Ultrasound-guided midline technique

INTERVENTIONS:
Other: Landmark technique — The site of needle insertion will be determined via manual palpation. A line joining the superior aspect of the iliac crests posteriorly (Tuffier's line') will be used as a surface landmark for the L4 vertebral body. The midline will be established by palpation of the tips of the spinous processes, and the site of needle insertion will be marked on the patient's skin. The interspace that appears widest, based on manual palpation, will be chosen for the first attempt. If the first attempt is unsuccessful, further attempts can be made at the same interspace or another interspace.
  Arms: Landmark technique
Other: Ultrasound-guided paramedian technique — The transducer will be applied in the parasagittal plane and the intervertebral levels will be identified by counting upwards from the sacrum (continuous hyperechoic line). The probe will then be angled obliquely to obtain a PSO view. The locations of the interlaminar spaces will be identified by visualizing the ligamentum flavum-dura mater complex and the posterior aspect of the vertebral body. The angulation at which the ligamentum flavum-dura mater complex and posterior vertebral body are best visualized will be considered the optimal angle for needle insertion and clearly communicated to the operator. The interlaminar space will be centered on the ultrasound screen and a skin marker will be used to make a mark on the patient's back at the middle of the ultrasound probe.
  Arms: Ultrasound-guided paramedian technique
Other: Ultrasound-guided midline technique — The transducer will be applied in the parasagittal plane, and after identification of the intervertebral levels, the probe will be rotated 90 degree to obtain the TM view. The transducer is moved in a cephalad-caudad direction between the spinous processes of L2 and L5 vertebra. The probe will be tilted slightly up and down to ensure a sufficient echogenic window at the selected intervertebral space. A skin marker will be used to make a mark on the patient's back at the middle of the ultrasound probe. The angle at which the ligamentum flavum-dura mater complex and the posterior aspect of the vertebral body are best visualized will be noted
  Arms: Ultrasound-guided midline technique

SUMMARY:
Traditionally, spinal anesthesia is performed using the palpation of bony landmark to identify the level and point of entry of the spinal needle. Recently, ultrasound imaging has become an increasingly popular procedure among anesthesiologists to guide neuraxial blockade. Most of the studies on pre-procedural ultrasound-guided neuraxial techniques are limited to a midline approach using a transverse median views. The parasagittal oblique view consistently offers better ultrasound view of the neuraxis compared to the transverse median view. However, it is still not evident whether these superior parasagittal oblique views will lead to an easier paramedian needle insertion. In the literature, there are no studies directly comparing the US-guided paramedian approach using the parasagittal oblique (PSO) view, the US-guided midline approach using the transverse median view, and the conventional landmark midline approach to perform spinal anesthesia in the elderly patients, in particular for the teaching of novice anesthesia residents.

DETAILED DESCRIPTION:
The aim of this study is to find out the optimal technique to perform spinal anesthesia by residents in training. Thus the investigators will compare preprocedural ultrasound-guided paramedian technique using parasagittal oblique view vs preprocedural ultrasound-guided midline technique using transverse median view vs landmark-guided midline technique of spinal anesthesia in the elderly population. Our hypothesis is that both preprocedural US-guided techniques are superior to the conventional landmark-guided midline technique with regard to ease of performance defined as success rate at first attempt, number of puncture attempts, spinal procedure time, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgery amenable to spinal anesthesia, aged more than 60 years, with American Society of Anesthesiologists physical status 1 to 4.

Exclusion Criteria:

* Patients who are unable to give consent, refuse spinal anesthesia, have spinal abnormalities (including scoliosis and previous spine operations with instrumentation) or have contraindications to spinal anesthesia, including allergy to local anesthetics or a bleeding diathesis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-11; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Rate of successful dural puncture on the first needle insertion attempt | up to 5 minutes from the start of insertion of the introducer of the spinal needle
  Rate of successful dural puncture on the first needle insertion attempt which is defined as the percentage of successful dural puncture on the first introducer needle advancement through skin; each skin puncture by introducer is considered as a needle insertion attempt.

SECONDARY OUTCOMES:
overall success rate in every technique | 60 minutes from the start of insertion of introducer of the spinal needle
  Overall success rate in every technique is defined as percentage of successful spinal anesthesia as evidenced by CSF flow through the spinal needle before spinal drug injection and a sensory block level >T10 15min after injection of spinal drug.
Number of introducer needle insertion attempts | 45 minutes from the start of insertion of introducer of the spinal needle
  Number of introducer needle insertion attempts is defined as the number of times the introducer needle was withdrawn from the skin and reinserted.
spinal procedure time | 60 minutes
  In groups US, period beginning when probe is first placed on patient's back and ending when examination is complete.
  In group LM, period beginning when patient's back is palpated first and ending when examination is complete.
patient satisfaction | 5 min after completion of administration of SA:
  Patient satisfaction will be scored as following:
  1. Very good
  2. Good
  3. Satisfactory
  4. Unpleasant
  5. Very unpleasant
Number of spinal needle redirections | 45 minutes
  Spinal needle redirected without complete withdrawal of the introducer of the spinal needle from skin

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Siddik-Sayyid, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rizk MS, Zeeni CA, Bouez JN, Bteich NJ, Sayyid SK, Alfahel WS, Siddik-Sayyid SM. Preprocedural ultrasound versus landmark techniques for spinal anesthesia performed by novice residents in elderly: a randomized controlled trial. BMC Anesthesiol. 2019 Nov 11;19(1):208. doi: 10.1186/s12871-019-0882-8. PMID 31711438